CLINICAL TRIAL: NCT00478530
Title: The Effect of Intravitreal Avastin on the Retina Measured by Electroretinogram
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Ygal Rotenstreich, Sheba Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-07-4573-YR-CTIL
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: ELECTRORETINOGRAM — Bevacizumab 1.25 mg/0.05 ml unilaterally into the vitreous cavity as part of the standard management for choroidal neovascular AMD. ERG responses form both eyes will be measured at baseline and 1 month after intravitreal injection

SUMMARY:
To evaluate the scotopic and photopic ERG responses before and after one month of intravitreal avastin injection in patients with choroidal neovascularization.

A positive finding that will reveal a toxic effect of intravitreal avastin injection on any component of the retina will have a significant important clinical impact regarding the decision whether the benefit of avastin treatment for CNV will prevail over toxic effect.

DETAILED DESCRIPTION:
The study will include 20 patients who are diagnosed with CNV and were submitted for intravitreal injection of avastin. Patients with uncontrolled glaucoma, any ocular operation two months prior to the injection, ocular inflammatory disease, systemic hypertension treated with more than one medication, myocardial infarct, congestive heart disease will not be included in the study. After the patient will approve to participate in the study and will fall in with the inclusion and exclusion criteria, the patient will sign a written consent statement (enclosed).

Medical history and ophthalmic examination will be written in the study file. The patients will undergo the full-field ERG test using the ISCEV Protocol. Since the ERG is a non invasive test the patient will be admitted on the same day for intravitreal avastin in the designated eye. After one month the patient will undergo identical ERG protocol in addition to the standard follow-up examinations protocol for intravitreal avastin injection (1 day, 1 week, 1 month). The other eye will serve as control group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were diagnosed with CNV caused by ARMD
2. ERG can be performed in both eyes

Exclusion Criteria:

1. Treatment within 7 days with VERTOPROFIN
2. Treatment within one month with laser photocoagulation
3. Ocular surgery for AMD (besides laser).
4. Participation in other medical study
5. Sub-fovea RPE atrophy in the study eye.
6. CNV with ocular histoplasmosis, trauma, pathological myopia.
7. Uveitis or history of uveitis.
8. Retinal pigment epithelium tear in the fovea of the injected eye.
9. Vitreous hemorrhage
10. Conjunctivitis, keratitis, scleritis, endophthalmitis.
11. Intraocular surgery (including cataract) within two months
12. Uncontrolled glaucoma (IOP≥30 mmHg under glaucoma medications)
13. Hypertension treated with two or more medication
14. History of myocardial infarct
15. History of myocardial insufficiency -

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-06 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
electroretinogram responses | before treatment and one month after treatment

CONTACTS AND LOCATIONS:
Overall Officials: YGAL ROTENSTREICH, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Background] Pai SA, Shetty R, Vijayan PB, Venkatasubramaniam G, Yadav NK, Shetty BK, Babu RB, Narayana KM. Clinical, anatomic, and electrophysiologic evaluation following intravitreal bevacizumab for macular edema in retinal vein occlusion. Am J Ophthalmol. 2007 Apr;143(4):601-6. doi: 10.1016/j.ajo.2006.12.037. Epub 2007 Feb 15. PMID 17306753
- [Derived] Rotenstreich Y, Harats D, Shaish A, Pras E, Belkin M. Treatment of a retinal dystrophy, fundus albipunctatus, with oral 9-cis-beta-carotene. Br J Ophthalmol. 2010 May;94(5):616-21. doi: 10.1136/bjo.2009.167049. Epub 2009 Dec 2. PMID 19955196